CLINICAL TRIAL: NCT05338476
Title: An Open-Label, Fixed-Sequence Study to Evaluate the Effect of Multiple Doses of LOXO-292 on the Single Dose Pharmacokinetics of Midazolam in Healthy Adult Subjects
Brief Title: A Study of Effects of Selpercatinib (LY3527723) on Midazolam in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 17753; J2G-OX-JZJR (Other: Eli Lilly and Company); LOXO-RET-18017 (Other: Loxo Oncology, Inc.)
Record Dates: First submitted 2022-04-19; First posted 2022-04-21 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1: Midazolam (Experimental): * Day 1: Participants received single oral dose of 2 milligram (mg) midazolam syrup.
  Interventions: Drug: Midazolam
- Period 2: Selpercatinib + Midazolam (Experimental): * Day 1 to Day 9: Participants received 160 mg Selpercatinib capsules twice daily (BID).
  * Day 10: Participant received 160 mg Selpercatinib capsules BID co-administered with a single oral dose of 2 mg midazolam syrup on the morning of Day 10.
  Interventions: Drug: Midazolam; Drug: Selpercatinib

INTERVENTIONS:
Drug: Midazolam — Administered orally.
Drug: Selpercatinib — Administered orally.
  Other Names: LY3527723; LOXO-292
  Arms: Period 2: Selpercatinib + Midazolam

SUMMARY:
The main purpose of this study is to assess the effect of selpercatinib on how fast midazolam gets into the blood stream and how long it takes the body to remove it when administered in healthy participants. Information about safety and tolerability will be collected. The study will last up to about 6 weeks, inclusive of screening period.

ELIGIBILITY:
Inclusion Criteria :

* Male and female participants of non-childbearing potential who are agreeable to take birth control measures until study completion
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per meter squared (kg/m²) and had a minimum weight of at least 50 kg at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), and blood and urine laboratory test results that are acceptable for the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Had blood loss of more than 500 milliliters (mL) within the previous 30 days of study screening
* Require treatment with inducers or inhibitors of cytochrome P450 (CYP) CYP3A within 14 days before the first dose of study drug through the end of Period 2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Period 1: Midazolam | Period 2: Selpercatinib + Midazolam
Started | 16 | 0
Safety Analysis Population (Received at Least One Dose of Study Drug) | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Period 1: Midazolam | Period 2: Selpercatinib + Midazolam
Started | 0 | 16 (Participants who completed Period 1, progressed to received treatment in Period 2.)
Safety Analysis Population (Received at Least One Dose of Study Drug) | 0 | 16 (1 participant discontinued the study after receiving the Selpercatinib dose on Day 5 in Period 2. Therefore, safety analysis population for Period 2: Selpercatinib + Midazolam (Day 10) treatment includes only the remaining 15 participants.)
Completed | 0 | 15
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: * Period 1: Participants received single oral dose of 2 milligram (mg) midazolam syrup on Day 1.
  * Period 2: Participants received 160 mg Selpercatinib capsules twice daily (BID) from Day 1-10, and on Day 10 it was co-administered with a single oral dose of 2 mg midazolam syrup on the morning of Day 10.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (6.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Last Observed Non-zero Concentration (AUC0-t) of Midazolam and Its Metabolite 1-hydroxymidazolam (1-OH-midazolam)
Description: PK: PK: AUC0-t of midazolam and its metabolite 1-OH-midazolam was reported.
Time Frame: Period 1: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 hours post dose); Period 2: Day 10 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- Period 2: Selpercatinib+ Midazolam: * Day 1 to Day 9: Participants received 160 mg Selpercatinib capsules twice daily (BID).
  * Day 10: Participant received 160 mg Selpercatinib capsules BID co-administered with a single oral dose of 2 mg midazolam syrup on the morning of Day 10.
Arm/Group | Period 1: Midazolam | Period 2: Selpercatinib+ Midazolam
Number analyzed (Participants) | 16 | 15
nanogram*hour per milliliter (ng*h/mL)
  Midazolam | 27.02 (38.4) | 42.43 (35.5)
  Metabolite: 1-OH-midazolam | 41.02 (100.7) | 55.81 (80.5)

2. Primary Outcome: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Midazolam and Its Metabolite 1-OH-midazolam
Description: PK: PK: AUC0-inf of midazolam and its metabolite 1-OH-midazolam was reported.
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Period 1: Midazolam | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16 | 15
nanogram*hour per milliliter (ng*h/mL)
  Midazolam | 28.46 (38.4) | 45.00 (36.7)
  Metabolite: 1-OH-midazolam | 43.29 (100.3) | 59.49 (80.2)

3. Primary Outcome: PK: Percent of AUC0-inf Extrapolated (AUC%Extrap) of Midazolam and Its Metabolite 1-OH-midazolam
Description: PK: PK: AUC%extrap of midazolam and its metabolite 1-OH-midazolam was reported.
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent AUC extrapolation
Arm/Group | Period 1: Midazolam | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16 | 15
percent AUC extrapolation
  Midazolam | 4.763 (36.9) | 5.165 (48.1)
  Metabolite: 1-OH-midazolam | 4.869 (41.3) | 5.849 (36.3)

4. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Midazolam and Its Metabolite 1-OH-midazolam
Description: PK: Cmax of midazolam and its metabolite 1-OH-midazolam was reported.
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Period 1: Midazolam | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16 | 15
nanogram per milliliter (ng/mL)
  Midazolam | 11.94 (32.0) | 16.76 (39.9)
  Metabolite: 1-OH-midazolam | 15.98 (70.1) | 17.91 (70.3)

5. Primary Outcome: PK: Time to Reach Maximum Observed Concentration (Tmax) of Midazolam and Its Metabolite 1-OH-midazolam
Description: PK: Tmax of midazolam and its metabolite 1-OH-midazolam was reported.
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Period 1: Midazolam | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16 | 15
hours
  Midazolam | 0.584 (20.4) | 0.626 (33.6)
  Metabolite: 1-OH-midazolam | 0.668 (25.3) | 0.738 (30.6)

6. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (Kel) of Midazolam and Its Metabolite 1-OH-midazolam
Description: PK: Kel of midazolam and its metabolite 1-OH-midazolam was reported.
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: One per hour (1/h)
Arm/Group | Period 1: Midazolam | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16 | 15
One per hour (1/h)
  Midazolam | 0.1193 (32.5) | 0.09787 (22.1)
  Metabolite: 1-OH-midazolam | 0.1105 (31.4) | 0.09474 (18.2)

7. Primary Outcome: PK: Apparent Terminal Elimination Half-life (t½) of Midazolam and Its Metabolite 1-OH-midazolam
Description: PK: t½ of midazolam and its metabolite 1-OH-midazolam was reported.
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Period 1: Midazolam | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16 | 15
hours
  Midazolam | 5.812 (32.5) | 7.082 (22.1)
  Metabolite: 1-OH-midazolam | 6.275 (31.4) | 7.317 (18.2)

8. Primary Outcome: PK: Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of Midazolam
Description: PK: CL/F of midazolam was reported.
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per Hour (L/h)
Arm/Group | Period 1: Midazolam | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16 | 15
Liter per Hour (L/h) | 70.26 (38.4) | 44.44 (36.7)

9. Primary Outcome: PK: Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) of Midazolam
Description: PK: Vz/F of midazolam was reported.
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Period 1: Midazolam | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16 | 15
Liter (L) | 589.1 (35.0) | 454.1 (32.3)

10. Secondary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 to the 12 Hour (AUC0-12) of Selpercatinib
Description: PK: AUC0-12 of Selpercatinib was reported.
Time Frame: Period 2: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16
ng*h/mL | 10710 (36.9)

11. Secondary Outcome: PK: Area Under the Concentration-time Curve During a Dosing Interval (Tau) at Steady State (AUCtau) of Selpercatinib
Description: PK: AUC0-tau of Selpercatinib was reported.
Time Frame: Period 2: Day 9 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose); Day 10 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 15
ng*h/mL
  Day 9 | 37610 (32.4)
  Day 10 | 36890 (33.5)

12. Secondary Outcome: PK: Maximum Observed Concentration (Cmax) of Selpercatinib
Description: PK: Cmax of Selpercatinib was reported.
Time Frame: Period 2: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16
ng/mL | 1859 (50.3)

13. Secondary Outcome: PK: Maximum Observed Concentration at Steady-state (Cmax,ss) of Selpercatinib
Description: PK: Cmax,ss of Selpercatinib was reported.
Time Frame: as for outcome 11
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 15
ng/mL
  Day 9 | 4574 (38.0)
  Day 10 | 4190 (36.8)

14. Secondary Outcome: PK: Concentration Observed at the End of the Dosing Interval (Ctrough) of Selpercatinib
Description: PK: Ctrough of Selpercatinib was reported.
Time Frame: Period 2: Predose at Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome. 'Number analyzed' signifies participants with available data at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16
ng/mL
  Day 1 | 1301 (23.1)
  Day 2 | 1843 (27.6)
  Day 3 | 2022 (29.4)
  Day 4 | 2213 (35.5)
  Day 5 | 2373 (34.9)
  Day 6: number analyzed (Participants) | 15
  Day 6 | 2660 (37.6)
  Day 7: number analyzed (Participants) | 15
  Day 7 | 2606 (32.7)
  Day 8: number analyzed (Participants) | 15
  Day 8 | 2733 (26.0)
  Day 9: number analyzed (Participants) | 15
  Day 9 | 2754 (30.9)

15. Secondary Outcome: PK: Time to Reach Maximum Observed Concentration (Tmax) of Selpercatinib
Description: PK: tmax of Selpercatinib was reported.
Time Frame: Period 2: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 16
hours | 1.843 (45.9)

16. Secondary Outcome: PK: Time to Reach Maximum Observed Concentration at Steady-state (Tmax,ss) of Selpercatinib
Description: PK: Tmax,ss of Selpercatinib was reported.
Time Frame: as for outcome 11
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 15
hours
  Day 9 | 1.955 (76.0)
  Day 10 | 1.752 (55.8)

17. Secondary Outcome: PK: Apparent Total Plasma Clearance at Steady State After Oral/Extravascular Administration (CL,ss/F) of Selpercatinib
Description: PK: CL,ss/F of Selpercatinib was reported.
Time Frame: as for outcome 11
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per Hours (L/h)
Arm/Group | Period 2: Selpercatinib + Midazolam
Number analyzed (Participants) | 11
Liter per Hours (L/h)
  Day 9 | 1.930 (35.8)
  Day 10: number analyzed (Participants) | 10
  Day 10 | 2.027 (34.5)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (up to Day 2 for Period 1; up to Day 11 for Period 2)
Description: Safety analysis population: All participants who received at least one dose of study drug.
  * 1 participant discontinued the study after receiving the Selpercatinib dose on Day 5 in Period 2. Therefore, safety analysis population for the Period 2: Selpercatinib + Midazolam (Day 10) treatment includes only the remaining 15 participants.
Groups:
- Period 1: Midazolam (Day 1): * Day 1: Participants received single oral dose of 2 milligram (mg) midazolam syrup.
- Period 2: Selpercatinib (Day 1 to Day 9): * Day 1 to Day 9: Participants received 160 mg Selpercatinib capsules twice daily (BID).
- Period 2: Selpercatinib + Midazolam (Day 10): * Day 10: Participant received 160 mg Selpercatinib capsules BID co-administered with a single oral dose of 2 mg midazolam syrup on the morning of Day 10.
Arm/Group | Period 1: Midazolam (Day 1) | Period 2: Selpercatinib (Day 1 to Day 9) | Period 2: Selpercatinib + Midazolam (Day 10)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 5/16 | 12/16 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Midazolam (Day 1) (N=16) | Period 2: Selpercatinib (Day 1 to Day 9) (N=16) | Period 2: Selpercatinib + Midazolam (Day 10) (N=15)
Hyperacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 4 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 8 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT05338476/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT05338476/SAP_001.pdf